CLINICAL TRIAL: NCT03568539
Title: An Open-label, Phase 1b Multicenter Study of IBI308 in Subjects With Advanced/Metastatic Solid Malignancies
Brief Title: IBI308 in Subjects With Advanced/Metastatic Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI308A102
Record Dates: First submitted 2018-05-01; First posted 2018-06-26 (Actual); Results first posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Advanced/Metastatic Solid Malignancies
Keywords: Advanced/metastatic solid malignancies, TMB high
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IBI308 (Experimental)
  Interventions: Drug: IBI308

INTERVENTIONS:
Drug: IBI308 — IBI308 200mg IV infusion, every 3 weeks.

SUMMARY:
The study is to evaluate preliminary anti-tumor activity (overall response rate, ORR) of IBI308 monotherapy in subjects with advanced/metastatic solid malignancies.

Patients will be recruited for 2 cohorts:

• Cohort 1: Advanced/metastatic cancers with TMB>10 mutations per megabase (mut/Mb). This enrollment of this cohort has been stopped per sponsor's communication with the sites. For patients who have already enrolled in this cohort, treatment and monitoring will be conducted as stipulated by the protocol. The patients will remain on study until disease progression or intolerable toxicity, death, withdrawal of consent, or end of study, whichever occurs first.

Cohort 2: Advanced/metastatic endometrial cancer (N=40)

ELIGIBILITY:
Inclusion Criteria:

1. Subjects able to give voluntary informed consent, understand the study and are willing to follow and complete all the test procedures.
2. Subjects (males and females) of childbearing potential should be willing to use reliable contraception methods that are deemed effective by the investigator from visit 1 through 90 days following the last dose of study drug. Postmenopausal women must have been amenorrhea for at least 12 months to be considered of non-childbearing potential.
3. Male or female subjects ≥18 years

   1. At least one measurable lesion (per RECIST version 1.1)
   2. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1.
   3. Subjects with life expectancy of ≥ 3 month
4. If subject received anti-tumor therapy:

   1. Generalized radiation therapy must have been completed 3 weeks prior to enrollment, or local radiotherapy or radiation therapy for bone metastases for 2 weeks prior to enrollment. Treatment with radiopharmaceuticals must have been completed 8 weeks prior to enrollment.
   2. Previous chemotherapy, biotherapy (tumor vaccines, cytokines, or growth factors that control cancer), tyrosine kinase inhibitors, or approved targeting and other treatments should have completed at least 3 weeks prior to the first administered dose in this study;
5. Subjects must have adequate organ function (liver, kidney function and hematopoietic function tests) prior IBI308 administration

   1. Absolute neutrophil count (ANC) ≥1.5 x10^9/L
   2. Platelet count ≥ 100 x 10^9/L
   3. Hemoglobin ≥ 9 g / dL (whole blood or component transfusion within 7 days before 1st dose of study drug is prohibited)
   4. Renal function tests: serum creatinine ≤1.5 ×upper limit of normal range (ULN) or an estimated glomerular filtration rate (eGFR) ≥ 50 mL/min/1.73 m2
   5. Liver function tests alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 x ULN, for patients with known liver cancer or liver metastases, AST and ALT ≤ 5 x ULN
   6. Total bilirubin (TBil) ≤1.5 x ULN; If Gilbert's Syndrome may have Bilirubin> 1.5 x ULN
   7. Coagulation tests: aPTT ≤ 1.5 x ULN and INR ≤2.0
6. Cohort Specific Inclusion Criteria:

Cohort 1: Advanced/metastatic cancers with high TMB expression

i. Advanced/metastatic cancers with TMB level > 10 mut/Mb ii. Histologically or cytologically confirmed unresectable Stage III/IV NSCLC or other advanced/metastatic cancers (for example, melanoma, bladder cancer, SCLC, prostate cancer, colorectal cancer, gastric cancer) iiI. Separate informed consent is required for subjects who provide fresh biopsies for serial tumor biopsies for biomarker testing. TMB testing should be performed on the most recently obtained tumor sample.

v. Subjects must be tested for TMB level before entering the study, and pre-screen informed consent is required for TMB testing. Subjects who have existing FoundationOne TMB testing results from within 6 months of study entry do not need to have repeat testing.

vi. Refractory or intolerant to standard therapy or for whom no standard therapy exists. Subjects must have no available therapy likely to confer clinical benefit for their cancer. Subjects who experienced irAE grade ≥ 3, or grade 2 recurrent pneumonitis, or who had to discontinue prior anti-PD-1/PD-L1 treatment due to irAEs of any grade will not be eligible.

vi. NSCLC subjects with EGFR mutation and/or ALK rearrangement and/or ROS-1 positive, should have received appropriate targeted therapy and are refractory to targeted therapy prior to enrolling this trial.

Cohort 2: Advanced/metastatic endometrial Cancer i. Histologically confirmed advanced/metastatic endometrial cancer. ii. Refractory or intolerant to standard therapy, and no available therapy likely to confer clinical benefit for their cancer. Subjects who experienced irAE grade ≥ 3, or who had to discontinue prior anti-PD-1/PD-L1 treatment due to irAEs of any grade will not be eligible.

Exclusion Criteria:

1. Legal incapacity or limited legal capacity.
2. Pregnancy, lactation, breastfeeding.
3. Concurrent anticancer treatment (e.g., cytoreductive therapy or cytokine therapy except for erythropoietin) or use of other investigational product within 28 days before start of trial treatment; major surgery within 28 days before start of trial treatment (excluding prior diagnostic biopsy.

   Note: Small molecule or antibody targeted therapy < 3 weeks from start of trial treatment will be excluded.
4. Received a biologic (G-CSF, GM-CSF) within 14 days prior to the first dose of study drug.
5. Vaccination within 4 weeks of first dose of IBI308 and while on study except for administration of inactivated vaccines (e.g., inactivated influenza vaccines)
6. Failure to recover from adverse events from the most recent anti-tumor treatment to CTCAE ≤ grade 1 or baseline with the exception of alopecia;
7. Active autoimmune disease requiring systemic treatment within the past 1 year or a documented history of clinically severe autoimmune disease or a syndrome that requires systemic steroids or immunosuppressive agents during the conduct of this study. Exceptions: - Vitiligo, eczema, psoriasis (<10% of body surface area (BSA) of skin eruption or systemic involvement) or resolved childhood asthma/atopy, autoimmune hypothyroidism stable on hormone replacement.
8. History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
9. Acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection.
10. History of primary immunodeficiency, stem cell or organ transplant, or previous clinical diagnosis of tuberculosis.
11. Subject who have had severe infection within 4 weeks or signs and symptoms of any active infection within 2 weeks prior to the first dose administration.
12. Known allergies, hypersensitivity, or intolerance to protein-based therapies or with a history of any significant drug allergy (e.g., anaphylaxis, hepatotoxicity, immune-mediated thrombocytopenia or anemia
13. Subjects who experienced (irAE) grade≥3 immunotherapy-related adverse events. Subjects with CNS metastasis unless they are asymptomatic or adequately treated with radiotherapy and/or surgery and subjects are neurologically stable with minimal residual symptoms/signs 14 days prior to dosing.
14. Patients who require high dose of systemic corticosteroids (>10 mg/day prednisone or equivalents) for at least 2 weeks prior to treatment are not eligible.
15. Severe or uncontrolled cardiac disease requiring treatment, congestive heart failure (New York Heart Association) NYHA III or IV, unstable angina pectoris even if medically controlled, history of myocardial infarction during the last 3 months, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia).
16. Any other serious underlying medical (e.g., uncontrolled hypertension, active uncontrolled infection, active gastric ulcer, uncontrolled seizures, cerebrovascular incidents, gastrointestinal bleeding, severe signs and symptoms of coagulation and clotting disorders, other serious cardiac conditions not listed in exclusion criteria), psychiatric, psychological, familial or geographical condition that, in the judgment of the investigator, may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2020-11-09 (Actual); Study Completion 2020-12-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - UC Irvine Medical Center, Orange, California
  - Northside Hospital, Inc, Atlanta, Georgia
  - Henry Ford Medical Center, Detroit, Michigan
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mary Crowley Cancer Research, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Final analysis data cutoff date: Dec20.
  39 subjects enrolled, 0 were ongoing.
Pre-assignment Details: 3 subjects on Cohort 1
  36 subjects on Cohort2
Groups:
- Cohort 1: Advanced/metastatic cancers with TMB>10 mutations per megabase (mut/Mb). 200mg IV Q3W.
- Cohort 2: Advanced/metastatic endometrial cancer. 200mg IV Q3W.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 3 | 36
Completed | 3 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 3 | 36 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 14 | 15
  >=65 years | 2 | 22 | 24
Age, Continuous [Median (Full Range); unit: Years] | 49.0 [44 to 78] | 67.5 [42 to 80] | 67.0 [42 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 36 | 38
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 4
  Not Hispanic or Latino | 3 | 31 | 34
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 2 | 28 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 36 | 39

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Confirmed)
Description: To evaluate preliminary anti-tumor activity (overall response rate, ORR) of IBI308 monotherapy in subjects with advanced/metastatic solid malignancies.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT/MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 29 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 34
Participants | 1 | 1

2. Secondary Outcome: Progression-free Survival
Description: To measure progression-free survival rate (PFS) Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non- target lesion, or the appearance of new lesions
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 34
Weeks | 17.14 [11.9 to 50.3] | 10.86 [5.7 to 12.0]

3. Secondary Outcome: Duration of Response
Description: To measure duration of response (DOR)
Time Frame: 2 years
Measure: Median (Full Range); unit: weeks
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 1 | 1
weeks | 46.14 [46.14 to 46.14] | 15.29 [15.29 to 15.29]

4. Secondary Outcome: Overall Survival
Description: To measure overall survival rate (OS)
Time Frame: 2 years
Population: A total of 37 subjects (3 subjects in Cohort 1 and 34 subjects in Cohort 2) were analyzed for efficacy in the full analysis set (FAS) population as 2 subjects in Cohort 2 were excluded from the FAS because they had no postbaseline tumor assessment of efficacy.
Measure: Median (95% Confidence Interval); unit: Week
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 34
Week | NA [50.3 to NA] — Median OS and OS range upper limit of 95% CI not reached | 61.86 [61.86 to NA] — OS range upper limit of 95% CI not reached

5. Secondary Outcome: Number of Participants With Detectable Anti- Drug Antibodies.
Description: Anti-Drug Antibodies will be tested to evaluate immunogenicity of IBI308
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 3 | 36
Participants | 0 | 1

6. Secondary Outcome: Area Under the Curve (AUC [0-504h])
Description: To evaluate the Area Under the Curve [AUC] of IBI308.
Time Frame: 0-504h
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*µg/mL
Groups:
- Cohort 1 & 2: intensive PK sampling set. 200mg IV Q3W.
Arm/Group | Cohort 1 & 2
Number analyzed (Participants) | 13
hr*µg/mL | 10400 (34.4)

7. Secondary Outcome: Maximum Plasma Concentration [Cmax]
Description: To evaluate the Maximum Plasma Concentration [Cmax] of IBI308.
Time Frame: Cycle 1 Day 1: predose, 5 minutes, 1, 6, 24, 48, 168, and 336 hr post-end of infusion
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Cohort 1 & 2
Number analyzed (Participants) | 13
µg/mL | 55.8 (18.5)

ADVERSE EVENTS:
Time Frame: 2 years
Description: Treatment-Emergent Adverse Events (TEAEs)
Groups:
- Cohort 2: Advanced/metastatic endometrial cancer 200mg IV Q3W.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 1/3 | 18/36
Serious Adverse Events (participants affected / at risk) | 2/3 | 12/36
Other Adverse Events (participants affected / at risk) | 3/3 | 34/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=36)
Urinary tract infection (Infections and infestations) | 0 | 3
Infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Gastrointestinal disorders) | 2 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal fistula (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=36)
Nausea (Gastrointestinal disorders) | 1 | 8
Diarrhoea (Gastrointestinal disorders) | 3 | 5
Abdominal pain (Gastrointestinal disorders) | 0 | 6
Abdominal distension (Gastrointestinal disorders) | 1 | 4
Vomiting (Gastrointestinal disorders) | 0 | 5
Constipation (Gastrointestinal disorders) | 0 | 3
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 15
Oedema peripheral (General disorders) | 2 | 6
Pyrexia (General disorders) | 1 | 2
Chills (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 3
Weight decreased (Investigations) | 0 | 4
Alanine aminotransferase increased (Investigations) | 1 | 1
Amylase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 6
Upper respiratory tract infection (Infections and infestations) | 0 | 3
Lung infection (Infections and infestations) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 3
Headache (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 2
Hot flush (Vascular disorders) | 1 | 2
Deep vein thrombosis (Vascular disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 5
Hypothyroidism (Endocrine disorders) | 0 | 4
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Haematuria (Renal and urinary disorders) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/39/NCT03568539/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT03568539/SAP_001.pdf